CLINICAL TRIAL: NCT07147270
Title: Impact of Patient Position on Chemical Pleurodesis by Chest Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, hieba gamal ezz-elragal awad, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU R107/2025
Record Dates: First submitted 2025-08-04; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Effect of Patient Rotation on Pleurodesis Success and Patient Comfort; Malignant Pleural Effusion; Pleurodesis
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no rotation after pleurodesis (No Intervention)
- rotation after pleurodesis (Active Comparator)
  Interventions: Other: side to side and front to back rotation 30 minutes each

INTERVENTIONS:
Other: side to side and front to back rotation 30 minutes each — side to side and front to back rotation 30 minutes each after pleurodesis
  Arms: rotation after pleurodesis

SUMMARY:
chemical pleurodesis using doxycycline is an acceptable and commonly employed palliation for malignant pleural effusion. Rotation of patient during pleurodesis using the powder from doxycycline capsule is still practiced in some centers. The benefit of rotation practice in pleurodesis can be verified after properly designed study on the outcome of pleurodesis with rotation and non-rotation by chest ultrasound assessment

DETAILED DESCRIPTION:
Pleurodesis through thoracoscopy could be done if the pleura appears abnormal on direct inspection thus offers diagnostic and therapeutic procedures in a single sitting. Talc is considered the best known sclerosing agent especially when used by medical thoracoscopy/pleuroscopy (MT/P). Unfortunately, a serious complication can occur with its use. Graded talc,which is the safest form is not available in many developing countries, including Egypt. Also, injectable tetracyclines' synthesis has been ceased worldwide.

Meanwhile, the oral forms of doxycycline are readily available, inexpensive and as effective as its parenteral forms in inducing pleurodesis. Therefore it will be used, aiming to assess the efficacy, safety and outcome of pleurodesis with and without patient rotation using doxycycline in malignant pleural effusion. Rotation of patients during tetracycline pleurodesis has been a common practice even at the moment. However, it had been proven that intrapleural instillation of parental tetracycline, a water soluble substance, to achieve chemical pleurodesis does not require rotation of patients as the tetracycline is distributed completely throughout the pleural space within seconds, and the distribution is not enhanced by patient's rotation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be admitted at Chest department, Ain-Shams University Hospitals with malignant pleural effusions candidate for pleurodesis

Exclusion Criteria:

* Multiloculated fluid
* Previous failed pleurodesis
* Liver failure
* Renal failure
* Congestive heart failure
* Prolonged use of steroids or NSAIDs
* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of pleural adhesion score in patients with malignant pleural effusion candidates for pleurodesis in group with rotation and the other without rotation | immediatly and after one month from pleurodesis
  study how patient rotation after pleurodesis affects its success by measuring pleural adherence score by chest ultrasound, a higher adhesion score means successful pleurodesis

SECONDARY OUTCOMES:
Measurement of non-verbal Pain score in patients with malignant pleural effusion candidates for pleurodesis in group with rotation and the other without rotation | immediately after pleurodesis
  Estimation of non-verbal pain score in patients with and without rotation after pleurodesis to assess how this rotation affects patients' comfort. A higher pain score means less comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
no participant data will be shared